CLINICAL TRIAL: NCT06318520
Title: Evaluation of the Clinical Success of Stainless Steel Crowns Applied Using Different Cements on Permanent Teeth Affected by Molar Incisor Hypomineralization
Brief Title: Clinical Success of Stainless Steel Crowns Applied Using Different Cements
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, Burcu Güçyetmez Topal, Asc. Prof., Afyonkarahisar Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AFSU-DHF-TOPAL-001
Record Dates: First submitted 2024-03-13; First posted 2024-03-19 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Dental Enamel Hypomineralization
Keywords: Dental Anomaly; Enamel; Stainless Steel Crowns
MeSH Terms: conditions — Dental Enamel Hypomineralization

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Calcium silicate based resin cement
  Interventions: Other: Use of Calcium silicate based resin cement and resin modified glass ionomer cement
- Arm 2 (Experimental): Resin modified glass ionomer cement
  Interventions: Other: Use of Calcium silicate based resin cement and resin modified glass ionomer cement

INTERVENTIONS:
Other: Use of Calcium silicate based resin cement and resin modified glass ionomer cement — Investigators will restore MIH teeth with stainless steel crowns using calcium silicate-based resin cement and resin-modified glass ionomer cement and evaluate their 1-year success.

SUMMARY:
The main question of the study was to evaluate the one-year clinical success of SSc bonded with two different cement types in MIH teeth with excessive material loss. The researchears will compare the survival rate, effect on gingival health and radiographic success of calcium silicate-based resin-containing cement and resin-modified glass ionomer cement.

DETAILED DESCRIPTION:
Molar incisor hypomineralization (MIH) is a developmental defect characterized by lack of mineralization in which one or more permanent first molars and often the incisors are also affected. In a study evaluating the prevalence of MIH in various countries, this rate was found to be 10%. It has been stated that it varies between 2.4-40. Its etiology is not known exactly, but it is thought to be due to reasons such as systemic, environmental and drug use encountered in the prenatal, perinatal and postnatal periods.

Molar incisor hypomineralization (MIH) is among the most important issues in pediatric dentistry today. Affected teeth show enamel opacities that range from white to brown depending on the duration of hypoplasia. Tooth brushing or tearing forces may cause posterior distortion, resulting in sensitivity. If dentin is exposed, resistance to tooth decay begins. Children with MIH require 10 times more treatment than normal. Although many studies can be done on etiological factors and prevalence, we are waiting for perspectives on the treatment of teeth affected by MIH. Deciding on the treatment method of teeth with MIH; the factors that produce the defect, whether the affected tooth is symptomatic or not, the age of the tooth and the expectations of the child/parent are taken into consideration. Although different restorative materials such as composite resins, glass ionomer cements or amalgam can be used in the care of these teeth, which are quite complex and difficult to treat, depending on the lesions, there is no consensus on the most effective treatment method. Since direct restorations are inadequate, especially in teeth with excessive material loss, the properties of materials that are resistant to fracture forces. Prefabricated stainless steel crowns (SSC), which have been preferred as the gold standard in long-term pediatric dentistry, are recommended for use in teeth affected by MIH. No study has been found in the accessible literature examining which bonding agent is more effective in the cementation of PCCs on teeth affected by MIH.

The aim of our study is to comparatively evaluate the 12-month clinical success of prefabricated stainless steel crowns cemented with calcium silicate-based adhesive resin cement or resin-modified glass ionomer cement on first molars diagnosed with MIH and with excessive material loss. In teeth affected by MIH, problems such as material loss, atypical restorations and sensitivity may be observed due to inorganic content and mineralization deficiency in the enamel tissue. It seems that these teeth do not last long and the treatments applied are not successful enough. It has been reported that the adhesion of restorative materials to the soft and hypomineralized enamel surface is low, therefore the risk of premature loss of restorations and secondary caries development is higher than that of healthy teeth. Therefore, stainless steel crowns are recommended as an alternative to direct restorations.

Many different materials can be used in the restoration of teeth with MIH; There are various factors affecting material selection. The severity of the defects, whether the affected tooth is symptomatic or not, the patient's dental age, the expected occlusal force for the restoration, the patient's risk of caries and oral hygiene status, and the child's/parent's expectations determine which restorative material will be used. For example; It was concluded that while conservative approaches are preferred in mild cases, the use of direct composite resin restorations, indirect restorations or metal crowns is a more appropriate treatment procedure in severe MIH cases. Restoration of teeth with MIH with SSC can prevent secondary caries, crown fractures and early tooth loss. One of the most important factors in the success of SSC is the cement material used. In recent years, self-hardening dual cure resin cements with their improved physical properties have been recommended for SSC bonding, and in vitro studies have clearly shown that they increase the success of restoration. However, no clinical study has been found in the literature showing how these cements affect the success of intraoral SSC in the long term. At the same time, although calcium silicate-based adhesive resin cements, which are a current material, have been used extensively in prosthetic studies, no study has been found in which they were used in SSC studies. One of the unique values of our study is that it is the first clinical study in which calcium silicate-based adhesive resin cements were used in SSC cementation. Another unique value is that it is the first study in which different cements were clinically compared for SSC bonding in teeth affected by MIH. We think that the results of our study will reduce the rate of recurrent treatment and therefore provide advantages to clinicians and families in terms of cost and time.

ELIGIBILITY:
Inclusion Criteria:

* Not having any systemic disease
* No history of allergy to any medication or restorative material (local anesthesia, nickel, etc.)
* No bad habits (mouth breathing, finger sucking, etc.)
* Score 3 or score 4 on the Frankl behavior scale
* Children between the ages of 9 and 12
* Agree to come to the controls regularly during the working period

Exclusion Criteria:

* Score 1 or 2 on the Frankl behavior scale
* Molar incisor hypomineralization has not been diagnosed
* Indication for unilateral crown
* Indication for extraction
* Gingival pocket depth exceeding 3 mm
* Presence of tooth mobility, abscess, fistula
* The opposite tooth of the affected tooth is absent or not in occlusion

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Anatomical Integrity | 3. month, 6. month, 9. month, 12. month
  0: The crown retains its anatomical integrity.
  1. The anatomical integrity of the restoration is impaired but functional.
  2. The restoration is fractured, displaced or completely lost.
Marginal Compliance | 3. month, 6. month, 9. month, 12. month
  0: Clinically ideal. No opening is observed between crown and gingiva, no sonde enters.
  1. Clinically acceptable. There is an opening between the crown and gingiva that does not extend to the prepared tooth.
  2. Clinically unacceptable, tooth mobility and an opening extending to the prepared tooth.
Proximal Contact | 3. month, 6. month, 9. month, 12. month
  0: Clinically ideal. It is possible to clean the proximal contact area with dental floss.
  1. Clinically acceptable. Floss passes hard or loose through the proximal contact area.
  2. Clinically unacceptable, proximal contact is not present.
Crown Marginal Location | 3. month, 6. month, 9. month, 12. month
  1. Subgingival
  2. Gingival level 3.Supragingival
Restoration success | 3. month, 6. month, 9. month, 12. month
  1. Crown appearance normal, no cracks, fractures, chips
  2. Inconspicuously small loss of material
  3. Huge loss of material
Green and Vermillion's Oral Hygiene Index | 3. month, 6. month, 9. month, 12. month
  0 No plaque and discoloration
  1. Plaque accumulation of less than 1/3 of the tooth surface or extrinsic staining without plaque accumulation and regardless of the surface covered
  2. Plaque accumulation more than 1/3 and less than 2/3 of the tooth surface
  3. Plaque accumulation covering more than 2/3 of the tooth surface

SECONDARY OUTCOMES:
Marginal Fit of the Crown (RADIOLOGICAL) | 6. month, 12. month
  1. There is no significant clearance between the crown and tooth surface.
  2. There is a significant clearance between the crown and the tooth surface.

CONTACTS AND LOCATIONS:
Overall Officials: Burcu GUCYETMEZ TOPAL, Asc. Prof., Study Director — Afyonkarahisar Health Sciences University; Esma ATIS, Res. Ass., Study Chair — Afyonkarahisar Health Sciences University
Locations (1):
- Afyonkarahisar Health Sciences University, Afyonkarahisar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No